CLINICAL TRIAL: NCT04304885
Title: Effect of Sonication on Periprosthetic Joint Infection Treatment Strategy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Orkhan Aliyev, Residents Doctor in Orthopedics Department, Bezmialem Vakif University
Other Study IDs: 28.02.2020-02
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Prosthesis-Related Infections; Hip Prosthesis Infection; Joint Infection; Biofilm
Keywords: total knee arthroplasty; complication; total hip arthroplasty; periprosthetic infection; revision arthroplasty; sonication; biofilm
MeSH Terms: conditions — Prosthesis-Related Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sonication method: The treatment strategies of all patients will be based on the cultural results to be made by the sonication method.
  Interventions: Diagnostic Test: Sonication method

INTERVENTIONS:
Diagnostic Test: Sonication method — Sonication dislodges adherent bacteria from explanted prosthetics by ultrasound and may improve the diagnosis of periprosthetic joint infection.

SUMMARY:
It is not known in the literature how much sonication affects the patient's treatment. Another important issue is that the place of this method in diagnosis is not clear. The aim of this study is to contribute to the literature on this issue and to determine the sensitivity and specificity of sonication prospectively using the new definition and effect of sonication on the treatment strategy in terms of infection in patients with PJI.

DETAILED DESCRIPTION:
Total knee and hip arthroplasties are successful surgical procedures that are widely applied all over the world and provide high patient satisfaction and increased quality of life. Periprosthetic joint infection (PJI), is a serious complication that negatively affects the targeted result, decreases patient satisfaction, and increases morbidity and mortality after total joint replacement. Another important issue, the previous infection is the most important reason for the failure of surgery in revision arthroplasty. It is known that the success of PJI treatment seriously can be affected by the type of microorganism and antibiotic sensitivity. Therefore, microbiological examination methods are always of interest, and one of them is the sonication method.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for revision arthroplasty (aseptic revision, septic revision, instability, and periprosthetic fracture)

Exclusion Criteria:

* who do not accept to participate in research
* insufficient data for new definition criteria
* acute periprosthetic infections
* patients with systemic inflammatory disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone primary hip and knee arthroplasty and will require revision for any reason.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-01-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 14 days
  To determine how many patients diagnosed with periprosthetic joint infection can be detected by sonication method.

SECONDARY OUTCOMES:
The change in antibiotic treatment. | 14 days
  In how many patients the sonication method will cause a change in treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Orkhan Aliyev, MD, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aliyev O, Yildiz F, Kaya HB, Aghazada A, Sumbul B, Citak M, Tuncay I. Sonication of explants enhances the diagnostic accuracy of synovial fluid and tissue cultures and can help determine the appropriate antibiotic therapy for prosthetic joint infections. Int Orthop. 2022 Mar;46(3):415-422. doi: 10.1007/s00264-021-05286-w. Epub 2022 Jan 24. PMID 35067748